CLINICAL TRIAL: NCT05579808
Title: The Effect of Epidural Analgesia on Labour and Neonatal and Maternal Outcomes in 1, 2a, 3, and 4a Robson's Classes: a Propensity Score-matched Analysis
Brief Title: Effect of Epidural Analgesia on Labour, Neonatal and Maternal Outcomes.
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 3741
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Labor Pain; Delivery Complication; Regional Anesthesia Morbidity
Keywords: Labor epidural analgesia
MeSH Terms: conditions — Labor Pain | interventions — Analgesia, Epidural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Epidural Analgesia
  Interventions: Procedure: Epidural Analgesia
- No analgesia

INTERVENTIONS:
Procedure: Epidural Analgesia — Using an aseptic technique while the patient is in sitting position, an epidural catheter was placed at the L2-L3 or L3-L4 interspace. Analgesia was established with the epidural administration of a low dose of local anaesthetic, plus a lipid-soluble opioid (ropivacaine 0.1% and sufentanyl 0.5%, 20 mL). Analgesia was maintained with a top-up regimen, using intermittent manual epidural boluses of increasing concentrations of ropivacaine, with up to 0.15% at full dilation, according to specific needs of individual participants.
  Groups: Epidural Analgesia

SUMMARY:
Lumbar epidural analgesia is the most used method for reducing labour pain, but its impact on the duration of the second stage of labour and on neonatal and maternal outcomes remains debated. The aim was of the study is to examine whether epidural analgesia affects the course and the outcomes of labour among patients divided according to the Robson-10 group classification system.

Patients of Robson's classes 1, 2a, 3, and 4a were divided into either the epidural analgesia group or the non-epidural analgesia group. A propensity score matching analysis was performed to balance intergroup differences. The primary goal was to analyse the duration of the second stage of labour. The secondary goals were to evaluate neonatal and maternal outcomes.

DETAILED DESCRIPTION:
Lumbar epidural analgesia (EA) is the recognized gold standard in labour pain control [1]. However, with data available to both support and refute a relationship between EA and a significant prolongation of the second stage of labour [1-4] (especially with low-dose anaesthetic protocols), its role is still controversial [5,6] . The second stage of labour is described as the period between complete cervical dilatation and the delivery of the baby. In 2014 the American College of Obstetricians and Gynecologists (ACOG) defined the normal duration of the second stage of labour as up to 2 hours in multiparous women and 3 hours in nulliparous ones [7]. However, as long as progress is being documented [7-9], newer recommendations propose longer durations based on individual factors [10,11] such as parity, maternal age [2] and body mass index (BMI) [12], hypertension [13], foetal weight and position [14], maternal position [15], oxytocin augmentation [2], and EA [16]. This study's attention on this phase of labour is strictly related to the potential impact of EA on foetal and maternal outcomes, and obstetric decision making [17-19]. In the literature, some papers report no detrimental foetal outcomes in cases involving a longer duration [3,20,21], while others show increased rates of maternal morbidity (third- or fourth-degree perineal lacerations, postpartum haemorrhage, and chorioamnionitis) [17,22] and Caesarean sections (CS), with labour dystocia as one of leading indications [19]. In order to investigate the effects of EA on labour effectively a propensity score matching seems appropriate. Propensity score matching is a statistical method for collecting data retrospectively that minimizes the selective biases that can arise from patients' backgrounds. Many studies have reported that propensity score matching produces results similar to RCTs despite its retrospective nature [4]. Based on five easily definable maternal characteristics, the Robson-10 classification system (RTGCS) introduced in 2001 and recognized by the WHO as the global standard for the analysis of pregnant patients [23], minimizes bias by comparing pregnant populations both within and across insitutions [24].

Using the propensity score matching method the present study aimed to analyse the impact of EA on the length of the second stage of labour and on foetal and maternal outcomes in the population of pregnant women referred to an Italian university hospital. These women have been stratified according to the RTGCS in order to settle the maternal characteristic confounders.

METHODS A retrospective cohort analysis was performed at a tertiary university hospital over an 11-year period (October 2008 to October 2019). This population was divided according to the RTGCS. Pregnant patients were enrolled according to the following RTGCS groups: R1 (nulliparous, single cephalic full-term pregnancy with spontaneous labour); R2a (nulliparous, single cephalic full-term pregnancy with induced labour); R3 (multiparous, single cephalic full-term pregnancy with spontaneous labour); and R4a (multiparous, single cephalic full-term pregnancy with induced labour). The exclusion criteria for this study were cases involving: multiple pregnancies, known major fetal or chromosomal abnormalities, pre-labour Caesarean deliveries, and elective Caesarean deliveries.

All maternal and obstetrical data were prospectively collected by labour and delivery unit personnel by entering cases into a perinatal database, which were then cross tabulated on an Excel file. The collected data included the demographic and obstetric parameters: maternal age and BMI, hypertension, diabetes, foetal weight and position, gestational age, labour induction (intravaginal or intracervical prostaglandin E2 gel, oxytocin), operative vaginal delivery (OVD) (only via the Kiwi OmniCup [produced by Clinical Innovations, Muray, Utah, USA] vacuum extractor), Caesarean section (CS), maternal morbidity (uterine atony, episiotomy, 3rd to 4th degree perineal laceration), and foetal morbidity (Apgar score< 7 at 1 and 5 minutes, neonatal resuscitation).

Access to EA is active on a 24-hour basis, with protocols reserving its administration for consenting women previously informed in an epidural outpatient clinic. All women who request analgesia for pain relief during labour are evaluated by an anaesthetist for suitability. Patients meeting absolute (i.e. uncorrected hypovolemia, coagulopathy, anticoagulant therapy) or relative (i.e. anatomical deformities, certain neurological disorders, sepsis) exclusion criteria are not qualified to receive EA. During labour, in the presence of a cervical dilatation of ≥3cm and in the active phase of the first stage (established by partograph), maternal status (blood pressure and temperature), and foetal well-being (20 minutes of normal cardiotocography) are also evaluated. In the absence of abnormalities, intravenous access by a 14-gauge (G) or 16G cannula is positioned and a crystalloid infusion is started. Using an aseptic technique while the patient is in sitting position, an epidural catheter is then placed at the L2-L3 or L3-L4 interspace. Finally, analgesia is established with the epidural administration of a low dose of local anaesthetic, plus a lipid-soluble opioid (ropivacaine 0.1% and sufentanyl 0.5%, 20 mL). Maternal blood pressure, foetal heart rate, pain scores, and the extent of sensory block are then assessed at five-minute intervals for the first 15 minutes, then at every half-hour. Analgesia is maintained with a top-up regimen, using intermittent manual epidural boluses of increasing concentrations of ropivacaine, with up to 0.15% at full dilation, according to specific needs of individual participants.

Statistical analysis As the use of observational data prevents the control of treatment assignment through randomization, systematic differences may be present between treated and untreated subjects in an randomized controlled trial. This can introduce confounding and thus prevent associations from being reliably estimated. However, the propensity score method is a statistical technique that aims to predict the probability of receiving treatment and/or having a condition based on identified covariates and background characteristics. Thus, the study population has been matched using a propensity score model with the optimal algorithm, including maternal age, BMI, gestational age, neonatal weight, parity, diabetes, and hypertension. The algorithm excluded patients with missing data in the matching variables. The quality of the matching was verified by considering an acceptable standard mean difference of <0.1 that was obtained in all participant groups. Data have been reported by mean ± standard deviation or by rate (i.e. percentage), unless indicated otherwise. All numerical variables with normal distributions were compared with t-tests, while categorical variables were compared with the chi-squared test or Fisher test when expected frequencies were less than 5. Statistical significance was considered for p-values <0.05. All analyses were performed in the R-statistical computing software 4.1.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women,
* at term (37-42 weeks),
* admitted to a tertiary university hospital over an 11-year period (October 2008 to October 2019)

Exclusion Criteria:

* multiple pregnancies,
* known major fetal or chromosomal abnormalities,
* pre-labour Caesarean deliveries,
* elective Caesarean deliveries.

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: A retrospective cohort analysis was performed of all live, at term (37-42 weeks) vaginal deliveries at a tertiary university hospital over an 11-year period (October 2008 to October 2019). This population was divided according to the RTGCS. Pregnant patients were enrolled according to the following RTGCS groups: R1 (nulliparous, single cephalic full-term pregnancy with spontaneous labour); R2a (nulliparous, single cephalic full-term pregnancy with induced labour); R3 (multiparous, single cephalic full-term pregnancy with spontaneous labour); and R4a (multiparous, single cephalic full-term pregnancy with induced labour).
Sampling Method: Non-Probability Sample
Enrollment: 21808 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Lenght of 2nd stage | From the time of the first documented full cervical dilatation to delivery
  Evaluate the length of the second stage of labour

SECONDARY OUTCOMES:
Foetal Outcome | At 1 and 5 minutes after birth
  Foetal outcome measured as Apgar's score
maternal outcome | 2 hours after the delivery.
  Incidence of uterine atony, 3rd and 4th degree lacerations, episiotomy, cesarean section and operative vaginal delivery.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico Agostino Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shen X, Li Y, Xu S, Wang N, Fan S, Qin X, Zhou C, Hess PE. Epidural Analgesia During the Second Stage of Labor: A Randomized Controlled Trial. Obstet Gynecol. 2017 Nov;130(5):1097-1103. doi: 10.1097/AOG.0000000000002306. PMID 29016499
- [Background] Ye Y, Song X, Liu L, Shi SQ, Garfield RE, Zhang G, Liu H. Effects of Patient-Controlled Epidural Analgesia on Uterine Electromyography During Spontaneous Onset of Labor in Term Nulliparous Women. Reprod Sci. 2015 Nov;22(11):1350-7. doi: 10.1177/1933719115578926. Epub 2015 Mar 29. PMID 25824008
- [Result] Anim-Somuah M, Smyth RM, Cyna AM, Cuthbert A. Epidural versus non-epidural or no analgesia for pain management in labour. Cochrane Database Syst Rev. 2018 May 21;5(5):CD000331. doi: 10.1002/14651858.CD000331.pub4. PMID 29781504
- [Result] Shmueli A, Salman L, Orbach-Zinger S, Aviram A, Hiersch L, Chen R, Gabbay-Benziv R. The impact of epidural analgesia on the duration of the second stage of labor. Birth. 2018 Dec;45(4):377-384. doi: 10.1111/birt.12355. Epub 2018 May 22. PMID 29790194
- [Result] Cheng YW, Shaffer BL, Nicholson JM, Caughey AB. Second stage of labor and epidural use: a larger effect than previously suggested. Obstet Gynecol. 2014 Mar;123(3):527-535. doi: 10.1097/AOG.0000000000000134. PMID 24499753
- [Result] Naito Y, Ida M, Yamamoto R, Tachibana K, Kinouchi K. The effect of labor epidural analgesia on labor, delivery, and neonatal outcomes: a propensity score-matched analysis in a single Japanese institute. JA Clin Rep. 2019 Jun 18;5(1):40. doi: 10.1186/s40981-019-0260-z. PMID 32026970
- [Result] Wang TT, Sun S, Huang SQ. Effects of Epidural Labor Analgesia With Low Concentrations of Local Anesthetics on Obstetric Outcomes: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Anesth Analg. 2017 May;124(5):1571-1580. doi: 10.1213/ANE.0000000000001709. PMID 27828798
- [Result] Obstetric care consensus no. 1: safe prevention of the primary cesarean delivery. Obstet Gynecol. 2014 Mar;123(3):693-711. doi: 10.1097/01.AOG.0000444441.04111.1d. PMID 24553167
- [Result] Zhang J, Landy HJ, Ware Branch D, Burkman R, Haberman S, Gregory KD, Hatjis CG, Ramirez MM, Bailit JL, Gonzalez-Quintero VH, Hibbard JU, Hoffman MK, Kominiarek M, Learman LA, Van Veldhuisen P, Troendle J, Reddy UM; Consortium on Safe Labor. Contemporary patterns of spontaneous labor with normal neonatal outcomes. Obstet Gynecol. 2010 Dec;116(6):1281-1287. doi: 10.1097/AOG.0b013e3181fdef6e. PMID 21099592
- [Result] Gimovsky AC, Berghella V. Randomized controlled trial of prolonged second stage: extending the time limit vs usual guidelines. Am J Obstet Gynecol. 2016 Mar;214(3):361.e1-6. doi: 10.1016/j.ajog.2015.12.042. PMID 26928148
- [Result] ACOG Committee Opinion No. 766: Approaches to Limit Intervention During Labor and Birth. Obstet Gynecol. 2019 Feb;133(2):e164-e173. doi: 10.1097/AOG.0000000000003074. PMID 30575638
- [Result] O'Connell MP, Hussain J, Maclennan FA, Lindow SW. Factors associated with a prolonged second state of labour--a case-controlled study of 364 nulliparous labours. J Obstet Gynaecol. 2003 May;23(3):255-7. doi: 10.1080/0144361031000098361. PMID 12850854
- [Result] Carlhall S, Kallen K, Blomberg M. Maternal body mass index and duration of labor. Eur J Obstet Gynecol Reprod Biol. 2013 Nov;171(1):49-53. doi: 10.1016/j.ejogrb.2013.08.021. Epub 2013 Aug 29. PMID 24041847
- [Result] Bregand-White JM, Kominiarek M, Hibbard JU Consortium On Safe L. OS030. Hypertension and labor duration: Does it take longer? Pregnancy Hypertens. 2012 Jul;2(3):192. doi: 10.1016/j.preghy.2012.04.031. Epub 2012 Jun 13. PMID 26105244
- [Result] Ghi T, Maroni E, Youssef A, Morselli-Labate AM, Paccapelo A, Montaguti E, Rizzo N, Pilu G. Sonographic pattern of fetal head descent: relationship with duration of active second stage of labor and occiput position at delivery. Ultrasound Obstet Gynecol. 2014 Jul;44(1):82-9. doi: 10.1002/uog.13324. Epub 2014 May 28. PMID 24496823
- [Result] Moraloglu O, Kansu-Celik H, Tasci Y, Karakaya BK, Yilmaz Y, Cakir E, Yakut HI. The influence of different maternal pushing positions on birth outcomes at the second stage of labor in nulliparous women. J Matern Fetal Neonatal Med. 2017 Jan;30(2):245-249. doi: 10.3109/14767058.2016.1169525. Epub 2016 Apr 19. PMID 27028537
- [Result] Cheng YW, Hopkins LM, Laros RK Jr, Caughey AB. Duration of the second stage of labor in multiparous women: maternal and neonatal outcomes. Am J Obstet Gynecol. 2007 Jun;196(6):585.e1-6. doi: 10.1016/j.ajog.2007.03.021. PMID 17547906
- [Result] Gimovsky AC, Guarente J, Berghella V. Prolonged second stage in nulliparous with epidurals: a systematic review. J Matern Fetal Neonatal Med. 2017 Feb;30(4):461-465. doi: 10.1080/14767058.2016.1174999. Epub 2016 May 5. PMID 27050812
- [Result] Bannister-Tyrrell M, Ford JB, Morris JM, Roberts CL. Epidural analgesia in labour and risk of caesarean delivery. Paediatr Perinat Epidemiol. 2014 Sep;28(5):400-11. doi: 10.1111/ppe.12139. Epub 2014 Jul 18. PMID 25040829
- [Result] Zha Y, Gong X, Yang C, Deng D, Feng L, Luo A, Wan L, Qiao F, Zeng W, Chen S, Wu Y, Han D, Liu H. Epidural analgesia during labor and its optimal initiation time-points: A real-world study on 400 Chinese nulliparas. Medicine (Baltimore). 2021 Mar 5;100(9):e24923. doi: 10.1097/MD.0000000000024923. PMID 33655955
- [Result] Ravelli ACJ, Eskes M, de Groot CJM, Abu-Hanna A, van der Post JAM. Intrapartum epidural analgesia and low Apgar score among singleton infants born at term: A propensity score matched study. Acta Obstet Gynecol Scand. 2020 Sep;99(9):1155-1162. doi: 10.1111/aogs.13837. Epub 2020 Mar 20. PMID 32142154
- [Result] Laughon SK, Berghella V, Reddy UM, Sundaram R, Lu Z, Hoffman MK. Neonatal and maternal outcomes with prolonged second stage of labor. Obstet Gynecol. 2014 Jul;124(1):57-67. doi: 10.1097/AOG.0000000000000278. PMID 24901265
- [Result] Robson MS. Can we reduce the caesarean section rate? Best Pract Res Clin Obstet Gynaecol. 2001 Feb;15(1):179-94. doi: 10.1053/beog.2000.0156. PMID 11359322
- [Result] Betran AP, Torloni MR, Zhang JJ, Gulmezoglu AM; WHO Working Group on Caesarean Section. WHO Statement on Caesarean Section Rates. BJOG. 2016 Apr;123(5):667-70. doi: 10.1111/1471-0528.13526. Epub 2015 Jul 22. No abstract available. PMID 26681211
- [Result] Wang Q, Zheng SX, Ni YF, Lu YY, Zhang B, Lian QQ, Hu MP. The effect of labor epidural analgesia on maternal-fetal outcomes: a retrospective cohort study. Arch Gynecol Obstet. 2018 Jul;298(1):89-96. doi: 10.1007/s00404-018-4777-6. Epub 2018 May 18. PMID 29777348
- [Result] La Camera G, La Via L, Murabito P, Pitino S, Dezio V, Interlandi A, Minardi C, Astuto M. Epidural analgesia during labour and stress markers in the newborn. J Obstet Gynaecol. 2021 Jul;41(5):690-692. doi: 10.1080/01443615.2020.1755621. Epub 2020 Jun 4. PMID 32496840
- [Result] de Barros Duarte L, Moises EC, Carvalho Cavalli R, Lanchote VL, Duarte G, da Cunha SP. Distribution of fentanyl in the placental intervillous space and in the different maternal and fetal compartments in term pregnant women. Eur J Clin Pharmacol. 2009 Aug;65(8):803-8. doi: 10.1007/s00228-009-0645-4. Epub 2009 Mar 28. PMID 19330322
- [Result] Zhang L, Xu C, Li Y. Impact of epidural labor analgesia using sufentanil combined with low-concentration ropivacaine on maternal and neonatal outcomes: a retrospective cohort study. BMC Anesthesiol. 2021 Sep 22;21(1):229. doi: 10.1186/s12871-021-01450-2. PMID 34551718
- [Result] Antonakou A, Papoutsis D. The Effect of Epidural Analgesia on the Delivery Outcome of Induced Labour: A Retrospective Case Series. Obstet Gynecol Int. 2016;2016:5740534. doi: 10.1155/2016/5740534. Epub 2016 Nov 20. PMID 27990163
- [Result] Srebnik N, Barkan O, Rottenstreich M, Ioscovich A, Farkash R, Rotshenker-Olshinka K, Samueloff A, Grisaru-Granovsky S. The impact of epidural analgesia on the mode of delivery in nulliparous women that attain the second stage of labor. J Matern Fetal Neonatal Med. 2020 Jul;33(14):2451-2458. doi: 10.1080/14767058.2018.1554045. Epub 2019 Jan 4. PMID 30608007
- [Result] Simic M, Cnattingius S, Petersson G, Sandstrom A, Stephansson O. Duration of second stage of labor and instrumental delivery as risk factors for severe perineal lacerations: population-based study. BMC Pregnancy Childbirth. 2017 Feb 21;17(1):72. doi: 10.1186/s12884-017-1251-6. PMID 28222704
- [Result] Fritel X, Schaal JP, Fauconnier A, Bertrand V, Levet C, Pigne A. Pelvic floor disorders 4 years after first delivery: a comparative study of restrictive versus systematic episiotomy. BJOG. 2008 Jan;115(2):247-52. doi: 10.1111/j.1471-0528.2007.01540.x. Epub 2007 Oct 25. PMID 17970794
- [Result] Webb DA, Culhane J. Hospital variation in episiotomy use and the risk of perineal trauma during childbirth. Birth. 2002 Jun;29(2):132-6. doi: 10.1046/j.1523-536x.2002.00173.x. PMID 12000414